CLINICAL TRIAL: NCT01955746
Title: Parent-sibling Tracing (PST) Linkage Based Analysis in the Family of More Than Two Members With Type 1 Diabetes in Taiwan for Novel HLA and Non-HLA Candidate Risk Alleles Detection
Brief Title: PST Linkage Based Analysis in the Family of More Than Two Members With Type 1 Diabetes in Taiwan
Acronym: PATT
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG3C1151
Record Dates: First submitted 2013-09-30; First posted 2013-10-07 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2013-09

CONDITIONS: The Genetic Variation of Type 1 Diabetes

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 DM

SUMMARY:
The purpose of this study is to explore the susceptible genes for Type 1 diabetes in Taiwan through the new genetic study methods.

DETAILED DESCRIPTION:
As an unclear autoimmune disorder, the pathogenesis of type 1 diabetes (T1D) remains elusive. Among all the methods for studying diseases pathophysiology, genetic approach has valuable capability as being both hypothesis-testing and hypothesis-generating. Although geo-epidemiological studies show relatively higher prevalence of T1D in Caucasians than in Asians, whether genetic factors identified in T1D of Caucasians are essential for T1D in Asians is not yet clarified. Although the human leukocyte antigen (HLA) genotype variants have been reported to be associated with T1D, the odds ratio (ORs) is relatively low in Taiwan as comparing with western countries, some families are indeed more than one child with T1D. However, the genetic linkage study in T1D is still limited in Taiwan that hampered the drug development or research in T1D. Therefore, we intend to explore the susceptible genes for T1D of Taiwan in this study, which will provide further researcher directions for this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes on the criteria of the American Diabetes Association with a very low C-peptide level (<0.35 ng/mL) with or without the experience of diabetic ketoacidosis.
2. The subjects whose four grandparents are of Chinese Han origin

Exclusion Criteria:

1. Patients with ages of onset more than 35 years are excluded.
2. The families having any member with known possible type 2 diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The family of more than one member with T1D
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Type 1 diabetes gene | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan